CLINICAL TRIAL: NCT02006342
Title: Effectiveness of Subcutaneous Glargine On The Time To Closure of The Anion Gap in Patients Presenting to the Emergency Department With Diabetic Keto-acidosis: A Pilot Study
Brief Title: Effectiveness of Subcutaneous Glargine On The Time To Closure of The Anion Gap in Patients Presenting to the Emergency Department With Diabetic Keto-acidosis
Acronym: GT-COG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Pratik B Doshi, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-12-0535
Record Dates: First submitted 2013-11-20; First posted 2013-12-10 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Diabetic Ketoacidosis
Keywords: Diabetes Mellitus; Diabetic Ketoacidosis; Insulin Glargine; Anion gap; Metabolic acidosis
MeSH Terms: conditions — Diabetic Ketoacidosis; Diabetes Mellitus; Acidosis | interventions — Insulin Glargine; Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Glargine plus Regular Insulin (Experimental): Patient's with Diabetic Ketoacidosis receiving standard of care treatment with regular insulin drip, IV fluids and close monitoring, with the addition of subcutaneous Insulin Glargine within 2 hours of diagnosis.
  Interventions: Drug: Insulin Glargine; Drug: Regular Insulin
- Control - Regular Insulin (Active Comparator): Patient's with Diabetic Ketoacidosis receiving standard of care treatment with regular insulin drip, IV fluids and close monitoring.
  Interventions: Drug: Regular Insulin

INTERVENTIONS:
Drug: Insulin Glargine
  Other Names: Lantus Insulin
  Arms: Insulin Glargine plus Regular Insulin
Drug: Regular Insulin

SUMMARY:
To determine if co-administration of subcutaneous (SQ)Insulin glargine in combination with intravenous (IV) insulin decreases the time to resolution of ketoacidosis and requirement for ICU admission compared to IV insulin with delayed administration of SQ glargine for the treatment of diabetic ketoacidosis (DKA).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Blood Glucose >200
* potential of hydrogen (pH) < 7.3
* Bicarbonate < 18
* Ketonemia or Ketonuria
* Anion Gap > or = 16

Exclusion Criteria:

* Age < 18 years
* Pregnant
* End state renal disease (ESRD)
* Prisoners
* Patients in shock or requiring emergency surgery
* Those unwilling to consent for the trial
* Allergic to Insulin Glargine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pratik B Doshi, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Lyndon B Johnson Hospital, Houston, Texas
  - Memorial Herman Hospital-Texas Medical Center, Houston, Texas

REFERENCES:
- [Background] Shankar V, Haque A, Churchwell KB, Russell W. Insulin glargine supplementation during early management phase of diabetic ketoacidosis in children. Intensive Care Med. 2007 Jul;33(7):1173-1178. doi: 10.1007/s00134-007-0674-3. Epub 2007 May 17. PMID 17508198
- [Result] Doshi P, Potter AJ, De Los Santos D, Banuelos R, Darger BF, Chathampally Y. Prospective randomized trial of insulin glargine in acute management of diabetic ketoacidosis in the emergency department: a pilot study. Acad Emerg Med. 2015 Jun;22(6):657-62. doi: 10.1111/acem.12673. Epub 2015 May 25. PMID 26013711

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Glargine Plus Regular Insulin: Patient's with Diabetic Ketoacidosis receiving standard of care treatment with regular insulin drip, IV fluids and close monitoring, with the addition of subcutaneous Insulin Glargine within 2 hours of diagnosis.
  Insulin Glargine
  Regular Insulin
- Control - Regular Insulin: Patient's with Diabetic Ketoacidosis receiving standard of care treatment with regular insulin drip, IV fluids and close monitoring.
  Regular Insulin
Period: Overall Study
Arm/Group | Insulin Glargine Plus Regular Insulin | Control - Regular Insulin
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: All who were enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine Plus Regular Insulin | Control - Regular Insulin | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38.5 [31.5 to 45.5] | 41.5 [29.0 to 50.5] | 41 [29 to 49.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 14 | 10 | 24
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Time to Anion Gap Closure
Description: Anion Gap is a measure of acidosis that results from decompensated Diabetes Mellitus. Acidosis is the result of the body being unable to utilize glucose for energy production and instead uses fatty acid metabolism resulting in ketone formation. Anion Gap is a surrogate measure for the level of ketones resulting in the excess acid production. Results reported are adjusted for initial anion gap, etiology of diabetic ketoacidosis, and comorbidities.
Time Frame: Participants monitored from hospital admission to discharge, an average of 4 days
Population: While one participant in the glargine group did not receive glargine, all who were enrolled were analyzed (intention to treat analysis).
Measure: Mean (Standard Error); unit: hours
Arm/Group | Insulin Glargine Plus Regular Insulin | Control - Regular Insulin
Number analyzed (Participants) | 20 | 20
hours | 10.2 (6.8) | 11.6 (6.4)

2. Secondary Outcome: Number of Participants Admitted to the ICU
Description: The goal was to determine if the amount of patients admitted to the ICU could be reduced by providing more efficient resolution of the critical condition which is the acidosis.
Time Frame: Participants followed for the duration of the Emergency Department stay, an expected average of 12 hours
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Insulin Glargine Plus Regular Insulin | Control - Regular Insulin
Number analyzed (Participants) | 20 | 20
participants | 6 | 4

3. Secondary Outcome: Intensive Care Unit Length of Stay
Description: Determine the amount of time patient is admitted to the intensive care unit with the goal of assessing if more efficient correction of the acidosis results in decreased time in the intensive care unit for the patients.
Time Frame: Participants monitored from hospital admission to discharge, an average of 4 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Insulin Glargine Plus Regular Insulin | Control - Regular Insulin
Number analyzed (Participants) | 20 | 20
days | 1.8 [1.6 to 1.9] | 1.2 [0.8 to 1.8]

4. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of stay was determined to assess whether a more efficient correction of the acidosis will result in decreased time that the patient is admitted to the hospital. Results reported are adjusted for age, hospital site, and etiology of diabetic ketoacidosis.
Time Frame: Participants monitored from hospital admission to discharge, an average of 4 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Insulin Glargine Plus Regular Insulin | Control - Regular Insulin
Number analyzed (Participants) | 20 | 20
days | 3.9 (3.4) | 4.6 (3.6)

5. Secondary Outcome: Number of Participants Who Developed Hypoglycemia
Description: To determine whether it is safe to administer both IV and subcutaneous insulin, it is important to assure that patient's glucose does not drop to critically low level and lead to adverse events. Hypoglycemia was defined as less than or equal to 60mg/dL during 24 hours after anion gap closure.
  Anion Gap is a measure of acidosis that results from decompensated Diabetes Mellitus. Acidosis is the result of the body being unable to utilize glucose for energy production and instead uses fatty acid metabolism resulting in ketone formation. Anion Gap is a surrogate measure for the level of ketones resulting in the excess acid production.
Time Frame: Participants monitored during the 24 hours after anion gap closure
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Insulin Glargine Plus Regular Insulin | Control - Regular Insulin
Number analyzed (Participants) | 20 | 20
participants | 2 | 3

ADVERSE EVENTS:
Time Frame: 24 hours after anion gap closure
Description: Participants were systematically assessed for hypoglycemia. Anion Gap is a measure of acidosis that results from decompensated Diabetes Mellitus. Acidosis is the result of the body being unable to utilize glucose for energy production and instead uses fatty acid metabolism resulting in ketone formation. Anion Gap is a surrogate measure for the level of ketones resulting in the excess acid production.
Arm/Group | Insulin Glargine Plus Regular Insulin | Control - Regular Insulin
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glargine Plus Regular Insulin (N=20) | Control - Regular Insulin (N=20)
hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
The study had a limited sample size; therefore, the results cannot definitively answer the research question. Also, because a convenience sample was used, there might be selection bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes